CLINICAL TRIAL: NCT06690164
Title: Study on the Effect of Atorvastatin Co-administered With Omeprazole on Statin Lactone (SEACOL)
Brief Title: Study on the Effect of Atorvastatin Co-administered With Omeprazole on Statin Lactone
Acronym: SEACOL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023/00947
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2024-11

CONDITIONS: Metabolite
Keywords: atorvastatin; atorvastatin lactone; omeprazole
MeSH Terms: interventions — Atorvastatin; Omeprazole

STUDY DESIGN:
Intervention Model Description: 2-arm, parallel group assignment: Arm 1: Atorvastatin 40mg + Omeprazole 20mg Arm 2: Atorvastatin 40mg onl
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm 1 (Experimental): Atorvastatin 40mg once a day + Omeprazole 20mg once a day, both drugs to be taken for 30 days.
  Interventions: Drug: Atorvastatin 40mg Tablet; Drug: Omeprazole 20mg Capsule
- Control arm 2 (Active Comparator): Atorvastatin 40mg once a day to be taken for 30 days.
  Interventions: Drug: Atorvastatin 40mg Tablet

INTERVENTIONS:
Drug: Atorvastatin 40mg Tablet — once a day for 30 days
Drug: Omeprazole 20mg Capsule — once a day for 30 days
  Arms: Intervention arm 1

SUMMARY:
This is a 2-arm, prospective, randomized, parallel-group, open-label, longitudinal study that lasts 30 days for each study participant. This study aims to investigate the effect of co-administration of Omeprazole with Atorvastatin versus Atorvastatin monotherapy on atorvastatin lactone level.

Primary endpoint: Higher statin lactone level in intervention arm after 30 days.

Secondary endpoints:

Higher hs-CRP in intervention arm Lipid panel Incidence of adverse drug side effects (e.g. muscle-related or elevated LFTs

DETAILED DESCRIPTION:
Description of study visits:

Pre-screening, consenting process, and screening procedures: Potential subjects will be identified through (i) direct advertisement such as posters to be put up around NUS / NUH, (ii) indirect - through word or mouth or snowballing. Participants who are interested will be interviewed over the phone by the study's Clinical Research Coordinator (CRC). During the telephone interview, participants will be given a brief description of the study design and procedures to be followed. If the participant is eligible, with their verbal agreement, arrangement will be made for participants to visit NUHS IMU (located in NUS MD6, level 7) for a screening and enrolment visit.

Informed consent: Informed consent will be taken by the PI. The study will be explained to the participant in detail. This will be performed in the privacy of a closed-door room. During the consenting process, the study will first be explained to the participants and ample time will be provided for participants to read through the informed consent form. Participants will also be (i) given opportunity to clarify any doubts before acknowledging the consent form; (ii) allowed to return home to discuss their participation with their family prior to consenting. Non-English speakers will have the English informed consent form with a short consent form in their language, so that participants can understand the purpose of this study and what is required of them. If the participant agrees to participate, the informed consent form will be signed by the PI and the participant, in the presence of a prescribed witness. In the event that the participant is illiterate, or a short consent form will be used, an impartial witness will be present instead. A copy of the informed consent will be kept by both the PI and the participant. Enrolled subjects will be updated in the Screening and Enrolment Log. Unselected subjects will be documented in the Pre-screening Log.

(c) Screening and baseline data collection: Participants who have signed the informed consent form will be assessed for eligibility to participate, based on the following assessments: (i) Demographic data; (ii) Medical and medication history; (iii) history of adverse drug reactions (if any). Participants will be interviewed directly to provide the above health information; medical records will not be assessed. Based on the collected data, approval for participation will be finalized by either the PI or Co-PI. Participants who are eligible for the study will be informed by the CRC and enrolled as a subject for the study.

(d) Blood draw: Post-fasting (8 hours) whole blood will be drawn twice. 18mL will be collected by ventipuncture each time, once at the time of recruitment (before intervention) and a second time on the second visit (T2) 30 days after the start of the intervention period. This amounts to a total of 36mL of blood collected throughout the study period. Blood will be drawn into EDTA vacutainers. All samples will be transferred from NUHS IMU to the PI's research laboratory (located in CDrum lab, NUS MD6, level 8). All the blood will be spun down to plasma. With an estimated plasma extraction efficiency of 45% via centrifugation, we expect to obtain about 8.1mL of plasma from 18mL of blood. The plasma will be aliquoted and stored in a -80 degrees Celsius freezer until analysis. For atorvastatin lactone metabolite profiling, a 1mL aliquot will be subjected to protein precipitation and used for analysis. Another 1mL aliquot will be used for high sensitivity c-reactive protein (hs-CRP) assays using the cobas c-111 machine. Another 3mL of plasma will be used for lipid panel profiling using cobas c-111 machine. The remaining plasma samples will be stored at -80 degrees Celsius for repeated analysis, if necessary.

Randomization and treatment allocation: The study will be open-label since the primary endpoint is an objective pharmacokinetic parameter. Treatment allocation between the Atorvastatin + Omeprazole and Atorvastatin only arms will be generated by a random allocation sequence using real-time web-based randomization system (IVRS) in a 1:1 ratio. The desired allocation ratio (1:1) can be achieved using permuted block randomization. Block randomization ensures balance between the 2 groups, in which the order of allocation is chosen at random at the beginning of the block. Block size will be determined by the study team member.

Intervention group 1: Atorvastatin 40mg/day + Omeprazole 20mg/day Control group: Atorvastatin 40mg/day. The investigators target to recruit 78 patients, of whom 39 patients will be assigned to each of the 2 treatment arms. The pharmacist will dispense the IP to the study participants. Each participant will be supplied 30 tablets of Atorvastatin and those in the intervention arm will receive an additional 30 capsules of Omeprazole during the trial. A total of 60 tablets / capsules will be dispensed to each participant in the intervention arm and 30 tablets to each participant in the control arm. An additional 5 surplus tablets / capsules of each drug will also be supplied to replace any damaged or missing tablets / capsules. Atorvastatin and Omeprazole will all be packaged and coded by the manufacturer. The pharmacist will be provided with the code list and will dispense the IP to each participant based on the unique subject ID for that participant. A CRC will provide a prescription on the day of the study visit and ensure that it is kept at the appropriate storage condition prior to administration.

ELIGIBILITY:
Inclusion Criteria:

* Males between 21 and 75 years old or females between 50 and 75 years old
* No contraindications to the use of Atorvastatin amp; Omeprazole.
* Ability to comply with study requirements eg administer Atorvastatin and Omeprazole once daily and return for follow-up 1 month later.
* Capable of understanding the study requirements and provide informed written consent to participate.
* Have not taken any statins or proton pump inhibitors in the past 30 days.

Exclusion Criteria:

* Women of child-bearing age (<50 years old)
* Pregnancy / Planning to conceive or breast-feeding
* Current or recent history of liver disease / renal impairment / myopathy / rhabdomyolysis
* Recent history of alcohol or drug abuse
* Concurrent use of other drugs that may interact with Atorvastatin, Omeprazole eg clopidogrel
* Acute infection or illness
* Allergy to any statins or proton pump inhibitors
* Medical condition(s) that might compromise safety or successful completion of study

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Higher statin lactone level in intervention arm after 30 days | 30 days
  Measure and compare statin lactone levels in intervention arm 1 and control arm 2

SECONDARY OUTCOMES:
Higher hs-CRP in intervention arm after 30 days | 30 days
  Measure and compare high sensitivity-c reactive protein in intervention arm 1 and control arm 2
Lipid panel | 30 days
  Measure and compare low density lipoprotein (LDL), high density lipoprotein (HDL), total cholesterol (TC), and triglycerides (TG) in intervention arm 1 and control arm 2
Incidence of adverse drug side effects | 30 days
  With administration of atorvastatin with or without omeprazole (specifically, to look out for unexplained muscle ache or weakness, yellowing of the skin or eye whites, and brownish urine)

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Singapore (NUS) MD6 Level 8, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be stored in a de-identified manner. If required by other researchers, it can be shared anonymously. Otherwise, IPD will be used in a collectively analysis manner and only the final analysis results will be shared.

DOCUMENTS (2):
  • Study Protocol (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT06690164/Prot_000.pdf
  • Informed Consent Form (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/64/NCT06690164/ICF_001.pdf